CLINICAL TRIAL: NCT01512212
Title: New Thyroid Fine Needle Biopsy Apparatus
Brief Title: New Thyroid Fine Needle Aspiration Biopsy Apparatus
Acronym: fnab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SB Istanbul Education and Research Hospital (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Erhan Aysan, MD Prof., SB Istanbul Education and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: thyroid.iiab
Record Dates: First submitted 2012-01-10; First posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Thyroid Cancer
Keywords: thyroid; fine; needle; aspiration; biopsy; new; technique
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Diseases | interventions — Biopsy; 1-fluoro-2-nitro-4-azidobenzene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- single group (No Intervention): FNAB will be perform first with standart technique and after with new FNAB apparatus
  Interventions: Procedure: biopsy

INTERVENTIONS:
Procedure: biopsy — fnab
  Other Names: fnab

SUMMARY:
Evaluation of the effectivity of the new thyroid fine needle aspiration biopsy (FNAB) apparatus of which patented from Turkish Patent Institute.

DETAILED DESCRIPTION:
The author group of this investigation produced a new thyroid fine needle aspiration biopsy (FNAB) apparatus and patented it from Turkish patent Institute. FNAB indicated nodular goitre patients are the subjects of this research. First, the investigators will perform standart FNAB after this procedure will perform FNAB with new apparatus. The investigators will evaluate the aspirates according to number of cells and malignity ratio of cells.

ELIGIBILITY:
Inclusion Criteria:

* fine needle aspiration biopsy indicated noduler goiter patients

Exclusion Criteria:

* diffuse goiter

Ages: 17 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
number of cells | 2
  number of aspirated cells will be compared

SECONDARY OUTCOMES:
type of cells | 2
  type (benign, suspect, malign) of cells will be compared

CONTACTS AND LOCATIONS:
Overall Officials: adnan yuksel, prof, Study Chair — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Marmara, Turkey (Türkiye)